CLINICAL TRIAL: NCT04466514
Title: A Phase 1, 3-Way Crossover Study to Evaluate the Effect of Food on Pharmacokinetics of ASTX029
Brief Title: A Phase 1 Study to Evaluate the Effect of Food on Pharmacokinetics of ASTX029
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ASTX029-11
Record Dates: First submitted 2020-07-08; First posted 2020-07-10 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — ASTX029

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A - Fasting (Experimental): Fasting conditions
  Interventions: Drug: ASTX029
- Treatment B - Fed (Experimental): High-fat/high-calorie breakfast
  Interventions: Drug: ASTX029
- Treatment C - Fed (Experimental): Low-fat/low-calorie breakfast
  Interventions: Drug: ASTX029

INTERVENTIONS:
Drug: ASTX029 — Form: tablet; Route of Administration: oral

SUMMARY:
Open-label, single dose, randomized, three-period, crossover design study to evaluate the effect of food on the bioavailability of a single oral dose of ASTX029 in healthy adult male and female participants.

Following a screening period of up to 28 days, eligible participants will be enrolled and randomized to receive a single treatment (A, B, C) in a random order, with each treatment separated by an approximate 5-day washout period. The duration of the study is expected to be approximately 42 days.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving informed consent and complying with study procedures.
2. Male or female, 18 to 45 years of age, inclusive, at date of consent.
3. Body mass index (BMI) ≥ 18.0 to ≤ 32.0 kg/m2 and total body weight > 50 kg (110 lbs.) at Screening.
4. All female participants must have a negative pregnancy test at Screening and at each Check-in Visit; and one of the following:

   1. Using a medically acceptable form of birth control for at least 1 month prior to first dose [e.g., hormonal contraceptives (oral, patch, injectable or vaginal ring), intrauterine device, or a double barrier method (e.g., diaphragm, cervical cap, oral, patch or vaginal hormonal contraceptive, condom, spermicide, or sponge)];
   2. Documented as surgically sterile by hysterectomy, bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal ligation/tubal occlusion) at least 6 months prior to the first dose;
   3. Postmenopausal (no menstruation for a minimum of 12 months and confirmed by follicle stimulating hormone (FSH) and estradiol at Screening).
5. Medically healthy based on medical history, vital sign measurements, clinical laboratory test results, and physical examination.
6. Non-smokers (including nicotine-containing products) for at least 6 continuous months prior to the first dose.
7. Be willing and able to consume all contents of the standardized breakfast (high-fat and low-fat) within 30 minutes prior to dosing.

Exclusion Criteria:

1. Females who are pregnant, lactating, or planning to become pregnant during the study.
2. Reported life-time history and/or recent evidence of alcohol or drug/substance abuse disorder.
3. Participants with reported history of hypersensitivity to ASTX029, or any component of the study drug formulation.
4. Participants who suffer from clinically significant systemic allergic disease or have a reported history of significant drug allergies, including, but not limited to, a history of anaphylactic reactions, or allergic reactions due to any drug leading to significant morbidity.
5. Participants who test positive at Screening for human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), or Hepatitis C virus (HCV) antibody.
6. Participants who test positive at Screening or at Check-in for alcohol and/or drugs of abuse.
7. Participants who donated ≥ 500 mL of blood within 56 days prior to the first dose of study drug or ≥ 50 mL and ≤ 499 mL of blood within 30 days or plasma (e.g. plasmapheresis) within 14 days prior to the first dose of study drug.
8. Screening 12-lead ECG with measurable QTc interval of ≥430 msec for males, ≥440 msec for females;
9. Reported history or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR) including:

   1. Presence or history of predisposing factors to RVO or CSR (e.g., glaucoma or ocular hypertension, diabetes mellitus) or,
   2. Visible retinal pathology as assessed by examination at screening that is considered a risk factor for RVO or CSR such as:
   3. Evidence of optic disc cupping or,
   4. Evidence of new visual field defects on automated perimetry.
10. Reported history of glaucoma or presence of any retinal diseases, including but not limited to, floaters, retinal detachment, macular degeneration, diabetic eye disease, retinitis pigmentosa.
11. Reported history or presence of hepatitis and/or hepatic dysfunction, based on subject medical history and clinical laboratory test results.
12. Evidence of renal dysfunction, including estimated glomerular filtration rate ≤60 mL/min.
13. Use of prescription or non-prescription drugs, dietary supplements, or herbal supplements at the time of Screening and within 14 days prior to the first dose of the study drug.
14. Participants who have a history of difficulty in donating blood or difficulty with phlebotomy procedures, and poor venous access.
15. Participants who have participated in another clinical trial within 30 days prior to the first study period.
16. Study staff or first-degree relative of study staff or the Sponsor directly involved in the study.
17. Any condition which in the opinion of Investigator would interfere with the subject's ability to provide informed consent, comply with study instructions, confound interpretation of study results, or endanger the subject if he or she took part in the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter Cmax | Predose to 72 hours postdose, up to Day 4
  Maximum plasma concentration
Pharmacokinetic parameter AUC(0-t) | Predose to 72 hours postdose, up to Day 4
  Area under the concentration versus time exposures calculated to the last measurable observation
Pharmacokinetic parameter AUC(0-∞) | Predose to 72 hours postdose, up to Day 4
  Area under the concentration versus time exposures extrapolated to infinity

SECONDARY OUTCOMES:
Pharmacokinetic parameter Tmax | Predose to 72 hours postdose, up to Day 4
  Time to reach maximum plasma concentration
Pharmacokinetic parameter t1/2 | Predose to 72 hours postdose, up to Day 4
  Elimination half-life
Pharmacokinetic parameter Kel | Predose to 72 hours postdose, up to Day 4
  Terminal elimination rate constant
Number of participants with Treatment-Emergent Adverse Events (TEAEs) | Up to Day 42

CONTACTS AND LOCATIONS:
Locations (1):
- Frontage Clinical Services, Secaucus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No